CLINICAL TRIAL: NCT04496115
Title: The Impact of Mindfulness on Prenatal Depression, Anxiety and Stress in Mothers at Risk of Preterm Delivery
Brief Title: Mindfulness in High Risk Pregnancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102522
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Stress; Anxiety; Depression; Mindfulness
Keywords: Mindfulness; Antepartum; High Risk Pregnancy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Experimental): Mindfulness training
  Interventions: Behavioral: Mindfulness
- Control (No Intervention): Standard of Care

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness training
  Arms: Mindfulness Intervention

SUMMARY:
Anxiety, depression and stress are common during pregnancy. These have been found to negatively impact mother and child outcomes. When anxiety, depression, and stress are present in pregnant women, it is therefore important to manage them to improve the outcome of the mother and her child.

Although pregnancy itself has been shown to increase anxiety, depression and stress, these issues are further elevated in high-risk pregnancy groups. Mothers at risk of preterm delivery (less than 37 weeks gestational age), have been found to have higher rates of depression, anxiety and stress compared to uncomplicated term pregnancies. In addition, anxiety, depression and stress symptoms themselves increase the risk for preterm delivery, creating a vicious cycle for this high-risk group.

Mindfulness is a tool that has been during pregnancy to reduce depression, anxiety, and stress. Many studies have found mindfulness to be an appropriate management option in normal term pregnancies.

To date, there have been no studies that have looked at Mindfulness as a tool for mothers admitted due to risk of preterm delivery. This study will explore the impact of teaching mindfulness skills to inpatient mothers at risk of preterm delivery and studying its effects on maternal depression, anxiety, and stress.

This study involves providing Mindfulness strategies during the mother's inpatient admission for the risk of preterm delivery for four consecutive weeks. Participants will be enrolled through informed consent. All participants will be given pre and post participation questionnaires to examine the impact of mindfulness on anxiety, depression and stress. The participants will also be encouraged to maintain a weekly mindfulness log. The results of this research may lead to future studies looking at the impact of mindfulness practice for high-risk pregnancies. This will also help open up the possibility of offering such courses for inpatient and outpatient high-risk pregnancies in the future.

DETAILED DESCRIPTION:
BACKGROUND

Anxiety and depression are two of the most common psychological symptoms that manifest in pregnant women. A recent systematic review found the prevalence of prenatal anxiety to be 18.2% in the first trimester, 19.1% in the second trimester and 24.6% in the third trimester. A separate systematic review found rates of depression in the prenatal period to be 16.4%. These symptoms have been found to negatively impact maternal health as well as fetal and childhood development. It is therefore imperative that anxiety and depression be assessed in all pregnant mothers and to further implement interventions to improve outcomes for both the mother and fetus.

Pregnant mothers with admission to an inpatient ward due to increased risk for preterm delivery have been found to experience elevated levels of anxiety, depression and stress compared to term pregnancies. Furthermore, increased anxiety and depression have been linked to the risk of preterm labor, creating a vicious cycle. A 2017 study that assessed anxiety and depression in a population of pregnant mothers at risk of preterm labor found 35.1% to have anxiety and 69.8% having depressive symptoms. By managing the psychological symptoms experienced in this cohort of pregnant mothers, the rationale is that the risks associated with them might be reduced, providing improved maternal and fetal outcomes.

There have been several studies that have assessed the benefits of mindfulness as a tool in reducing anxiety, stress and depression specifically in pregnancy. A 2016 meta-analysis found that mindfulness-based interventions are effective at reducing pregnancy related depression, stress, and anxiety. A randomized controlled trial assessed pregnant women with high levels of stress and anxiety after six weeks of mindfulness practice with results demonstrating larger decreases in pregnancy specific anxiety as compared to the control group.

Mindfulness has been implemented as an intervention prior to delivery with encouraging results. It has also been used in the post-partum period in environments such as the Neonatal Intensive Care Unit (NICU), where parental anxiety, depression and stress are elevated due to admission of their newborn after birth. Recent studies have shown that when mindfulness is used in the NICU environment, it assists with reduction of depressive, anxiety and trauma symptoms as well as improving maternal sleep Mindfulness also helped mothers deal with acute stressors more appropriately and promoted awareness and reduced stress related emotions.

To date, there have been no studies that have looked at Mindfulness as a tool for mothers admitted due to risk of preterm delivery. The study being proposed here, would assess the impact of mindfulness in the prenatal period, in a group of mothers who are experiencing elevated levels of depression, anxiety and stress due to the risk of preterm delivery.

HYPOTHESIS

The investigators hypothesize that pregnant women will experience less depression, anxiety and stress with mindfulness and will increase their mindful awareness.

MATERIALS AND METHODS

This study is a non blinded, prospective randomized controlled trial.

Following recruitment of participants, randomization into either the mindfulness group or the control group will occur.

Mindfulness Group (MG)

Participants within the mindfulness group will be instructed by a mindfulness practitioner/coach once a week for four weeks in one-on-one sessions. Weekly journals will be provided to measure adherence. Optional mindfulness audio files may be used to continue mindfulness practice in between guided mindfulness sessions.

Control Group (CG)

Participants within the control group will receive care as usual without any additional mindfulness techniques provided during the four-week period.

Instruments

* General Demographic Form: A researcher created maternal demographic data form (age, educational level, number of gestations, parity, prior experience with mindfulness, history of depression and anxiety) to be completed by the mother at enrolment.
* Depression, Anxiety and Stress Scale: 21 item Depression, Anxiety, Stress Scale to be completed by the mother at enrolment and at the end of the four weeks.
* Pregnancy Related Anxiety Scale: 10 item Pregnancy Related Anxiety Scale to be completed by the mother at enrolment and at the end of the four weeks.
* Mindfulness Scales: 15 item Mindfulness Attention Awareness Scale and the 13 item Toronto Mindfulness Scale will be completed by the mother at enrolment and at the end of the four weeks.
* Mindfulness Weekly Journal: Document recording the duration of mindfulness practice every day during the four-week intervention to assess adherence.

COVID-19 info

There will be in-person recruitment and data collection, but all in-person interactions will be put on hold until social distancing requirements have been lifted.

DATA ANALYSIS

Study data will be managed using Research Electronic Data Capture, a secure, web-based software platform, hosted at the University of Alberta. Group demographics were compared with t-test, chi-square and Mann-Whitney U as appropriate. The scores of the four questionnaires will be analyzed with the Wilcoxon Signed-Rank test for within group comparison and the Mann-Whitney U test for between group comparisons. The Spearman correlation test will be used in the mindfulness group for correlation between the mindfulness scores and the stress, anxiety and depression scores. 2-tailed p-values will be used.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers admitted to the antepartum ward at the Lois Hole Hospital for risk of preterm delivery (< 34 weeks GA) are eligible for the study.
* if they speak, read and write English,
* if their inpatient stay is anticipated to be at least 4 weeks following recruitment
* if they are willing and able to attend the mindfulness sessions.

Exclusion Criteria:

* if they are experiencing current mental illness issues
* if they are experiencing current or prior substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in stress symptoms | Change from recruitment to 4 weeks after
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of stress symptoms. Minimum score is 0. Maximum score is 21.
Change in anxiety symptoms | Change from recruitment to 4 weeks after
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). Minimum score is 0. Maximum score is 21.
  And using the Pregnancy Related Anxiety Scale. Scores for individual question range from 1 (Not at all) to 5 (Very much). Minimum score is 10. Maximum score is 50.
  A high score in both scales means a high level of anxiety symptoms.
Change in depression symptoms | Change from recruitment to 4 weeks after
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of depression symptoms. Minimum score is 0. Maximum score is 21.
Change in mindful awareness | Change from recruitment to 4 weeks after
  using the Mindfulness Attention Awareness Scale. Scores for individual question range from 1 (Almost Never) to 6 (Almost Always). Minimum score is 15. Maximum score is 90.
  And using Toronto Mindfulness Scale. Scores for individual question range from 0 (Not at all) to 4 (Very much). This scale has 2 subscales. Minimum score is 0. Maximum score is 24 for the first subscale and 28 for the second subscale.
  A high score in both scales (and subscales)means a high mindful awareness level.

SECONDARY OUTCOMES:
Mindfulness practice | 4 weeks
  Duration of mindfulness practice
Gestational age | variable (less than 20 weeks from recruitment)
  Gestational age of the newborn (in weeks and days) at the time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine Landry, MD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No